CLINICAL TRIAL: NCT06367010
Title: Clinical Efficacy and Safety Analysis of 125I Brachytherapy Combined With Anlotinib in Radioiodine Refractory Thyroid Carcinoma Patients
Brief Title: Clinical Efficacy of 125I Brachytherapy Combined With Anlotinib in Radioiodine Refractory Thyroid Carcinoma Patients
Status: Completed | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-36-24-010942
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Neoplasms
Keywords: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms | interventions — anlotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Iodine-125 brachytherapy combine with Anlotinib — Iodine-125 brachytherapy combine with Anlotinib

SUMMARY:
A retrospective analysis was conducted on patients with radioiodine-refractory thyroid carcinoma (RRTC) who underwent radioactive 125I seed implantation combined with anlotinib from January 2019 to October 2024 at Jiangxi Cancer Hospital. Data on tumor size changes before and after treatment, serological tests (including serum TG, TgAb, CTn, CEA, etc.), changes in patients' pain scores, and side effects were collected to evaluate the clinical efficacy and safety of this therapy.

DETAILED DESCRIPTION:
A retrospective analysis was conducted on RRTC patients who underwent radioactive 125I seed implantation combined with anlotinib from 2019 to 2024 at Jiangxi Cancer Hospital, including 2 cases of papillary thyroid carcinoma (PTC), 4 cases of follicular thyroid carcinoma (FTC), and 2 cases of medullary thyroid carcinoma (MTC).

Prior to the treatment, patients were informed about their condition, the expected efficacy, and the potential side effects and toxic effects of 125I seed implantation therapy combined with anlotinib. All patients accepted the treatment plan and signed an informed consent form. The preoperative evaluation process includes assessments of coagulation function, liver and kidney function, cardiopulmonary function, and local CT scans.

A collaborative effort between physicians and physicists was undertaken to establish a treatment regimen with a prescription dose ranging from 80 to 120 Gy. The CT-guided 125I seed implantation procedure was conducted according to the prescribed treatment regimen. On the day of completion of the 125I seed implantation procedure, all patients began treatment with anlotinib. Patients undergo 14 consecutive days of treatment followed by 7 days off, constituting one cycle. This cycle is repeated until progressive disease (PD) occurs or the patient shows intolerance to the treatment.

Subsequent evaluations were scheduled post-surgery, focusing on lesion dimensions, serum Tg levels, pain levels, and adverse reactions. Lesion size was determined using CT imaging. Each measurable lesion underwent an average measurement derived from a minimum of three readings, with all measurements conducted by the same individual to minimize measurement discrepancies.

Response Evaluation Criteria in Solid Tumors (RECIST 1.1) [1] were used to assess treatment response. Use the Visual Analogue Scale to record patients' pain scores. Adverse reactions, including infection, bleeding, pneumothorax, bone marrow suppression, and seed displacement, were recorded. Adverse events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.The data were analyzed using IBM SPSS 27.0.

ELIGIBILITY:
Inclusion Criteria:

* (i) Thyroid cancer confirmed through pathological examination;
* (ii) Disease progression after conventional treatments, such as surgery, postoperative 131I, and external irradiation;
* (iii) Multiple tumor foci, with at least one focus where the tumor's maximum diameter exceeds 3 cm.

Exclusion Criteria:

* (i) Patients who are positive for TgAb;
* (ii) Patients with a TSH level of 0.1 mU/L or higher;
* (iii) Patients with severe coagulation disorders;
* (iv) Patients with severe cardiorespiratory impairment;
* (v) Patients who are unable to cooperate with or tolerate particle implantation surgery;
* (vi) Patients with an expected survival period of less than 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with radioiodine-refractory thyroid carcinoma can receive a radioactive 125I particle treatment combined with anilotinib.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The CT images were used to measure the change in the maximum diameter of the lesion in millimeters. | Patients were evaluated preoperatively and at 2, 4, and 6 months postoperatively.
  Lymph nodes were assessed based on their shortest diameter, while other target lesions were evaluated based on their longest diameter. Each measurable lesion underwent an average measurement derived from a minimum of three readings, with all measurements conducted by the same individual to minimize measurement discrepancies. Response Evaluation Criteria in Solid Tumors (RECIST 1.1) were used to assess treatment response[1].
Serological assessment | Patients were evaluated preoperatively and at 2, 4, and 6 months postoperatively.
  Including serum Thyroglobulin (Tg) and serum Anti-thyroglobulin Antibody levels (TgAb) in thyrotropin-inhibited states, as well as tumor markers such as Carcinoembryonic Antigen (CEA).
Use the Numerical Rating Scale (NRS) to record patients' pain scores. | Patients were evaluated preoperatively and at 2, 4, and 6 months postoperatively.
  The scale ranges from 0 to 10 points, with pain increasing incrementally. 0 indicates no pain, 1-3 indicate mild pain that is still tolerable and does not interfere with sleep or normal life, 4-6 indicate moderate pain that interferes with sleep and requires analgesic medication to alleviate it, and 7-10 show intense and intolerable pain that seriously interferes with sleep and diet and requires strong analgesic drugs.
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Assess within six months after surgery.
  Adverse reactions, such as pain, pneumothorax, hemorrhage, myelosuppression, infection, radiation inflammation, necrosis, hand-foot syndrome, hypertension, proteinuria, and diarrhea, were observed and recorded. The severity of the adverse reactions was graded according to the CTCAE v5.0, with grades ranging from 1 to 5, where grade 1 represents the mildest and grade 5 the most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Chen, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe H, Okada M, Kaji Y, Satouchi M, Sato Y, Yamabe Y, Onaya H, Endo M, Sone M, Arai Y. [New response evaluation criteria in solid tumours-revised RECIST guideline (version 1.1)]. Gan To Kagaku Ryoho. 2009 Dec;36(13):2495-501. Japanese. PMID 20009446